CLINICAL TRIAL: NCT05344352
Title: Studio Clinico Randomizzato in Doppio Cieco, Controllato Verso Placebo, a Gruppi Paralleli Sull'efficacia Clinica Di Un Prodotto a Base Di Probiotici Nel Migliorare I Sintomi Della Rinite Allergica Perenne E Stagionale
Brief Title: Effect of a Multistrain Probiotic on Allergic Rhinitis Symptoms and Gut Microbiota Composition in Atopic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Giacomo Caio, Professor, MD, PhD, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AllergAway2021
Record Dates: First submitted 2022-03-30; First posted 2022-04-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2023-05

CONDITIONS: Allergic Rhinitis
Keywords: Microbiota
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mutistrain probiotic (Active Comparator)
  Interventions: Dietary Supplement: Multistrain Probiotic
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Multistrain Probiotic — 8-week daily administration
  Arms: Mutistrain probiotic
Other: Placebo — 8-week daily administration
  Arms: Placebo

SUMMARY:
The purpose of the current study is to evaluate the efficacy of administering a multistrain probiotic in adult human subjects suffering from allergic rhinitis and evaluate both symptomatology through validated questionnaires and gut microbiota modification during and after treatment.

DETAILED DESCRIPTION:
Adult subjects (18-60) with documented allergic rhinitis will be assigned to placebo or probiotic groups and take either placebo or probiotic dietary intervention for 8 weeks. Total nasal symptom score (TNSS), Rhinitis Control Assessment Test (RCAT), Mini Rhinoconjunctivitis Quality of Life Questionnaire (MiniRQLQ) will be compared over 12 weeks between the two treatment groups. In addition, serological markers (Eosinophil count, Total IgE and Eosinophilic cationic protein) and gut microbiota features will be evaluated over a 12 week period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years of age
* Established allergic rhinitis (clinical history of rhinorrhea, congestion, sneezing, pruritis >2 years)
* Positive Skin Prick Test and/or Specific IgE to at least one aeroallergen.
* Have signed the consent form
* Have been instructed during screening and agreed to not take any probiotic containing products outside the study for the study period

Exclusion Criteria:

* Subjects currently under treatment with antibiotics
* Subjects undergoing allergen immunotherapy
* Pregnancy
* Vasomotor rhinitis
* Nasal cavity disorders
* Ear infections
* Other chronic diseases (e.g. gastrointestinal, cardiovascular, infections)
* Subjects diagnosed with non-controlled asthma
* Subjects currently participating in another interventional clinical trial or having participated in another clinical trial in the last 2 months
* Subjects on chronic use of systemic corticosteroids
* Proton pump inhibitors 2-weeks prior to randomization
* Antibiotics 2-weeks prior to randomization

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Total nasal symptom score (TNSS) | over 8 weeks + 4 week after the end of trial (follow-up)
  Total nasal symptom score (TNSS) measuring nasal congestion, runny nose, nasal itching and sneezing on a scale of 0-12 will be compared over 8 weeks between the two treatment groups + after 4 weeks from the end of trial.

SECONDARY OUTCOMES:
Rhinitis Control Assessment Test (RCAT) | over 8 weeks + 4 week after the end of trial (follow-up)
Mini Rhinoconjunctivitis Quality of Life Questionnaire (MiniRQLQ) | over 8 weeks + 4 week after the end of trial (follow-up)
Gut Microbiota changes on fecal samples | over 8 weeks + 4 week after the end of trial (follow-up)
  Shotgun metagenomic sequencing and computational profiling with the tools in bioBAkery3. MetaPhlAn3.0 and HUMAnN3.0 will be used for taxonomic and functional profiling. Only the species showing a non-zero abundance in ≥5% of the samples will be considered in the cross-sectional and longitudinal analysis. P-values will be corrected for multiple hypothesis testing with Benjamini-Hochberg FDR procedure, and the longitudinal analysis was performed using a linear mixed-effects model.
Serological markers | over 8 weeks + 4 week after the end of trial (follow-up)
  ECP, Eosinophil count, total IgE

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria di Ferrara, Cona, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No